CLINICAL TRIAL: NCT01394146
Title: Impact of Food Additives on Phosphorus Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Orlando M. Gutierrez, MD, MMSc, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: F110118001
Record Dates: First submitted 2011-07-12; First posted 2011-07-14 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: phosphorus-based food additives; phosphorus metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects with healthy kidney function (Experimental)
  Interventions: Other: Research diet

INTERVENTIONS:
Other: Research diet — Participants will be provided specially prepared meals to eat at home for two weeks. During the first week, participants will eat foods that do not have any phosphorus-based food additives in them (this is called the control diet). During the second week, participants will eat foods that all have phosphorus-based food additives in them (called the intervention diet).

SUMMARY:
The purpose of the study is to learn more about how phosphorus-based food additives affect phosphorus metabolism in people with normal kidney function.

DETAILED DESCRIPTION:
Phosphorus is a mineral that is found in foods such as dairy products, nuts, and meat, and is important for strengthening the bones. However, too much phosphorus in the blood may be bad for the health of your heart and blood vessels. The kidneys keep the blood levels of phosphorus normal by getting rid of extra phosphorus in the urine. New research has found that common forms of food additives that are high in phosphorus may increase blood phosphorus levels in individuals with kidney disease. In addition, these food additives may increase blood levels of hormones that control phosphorus such as parathyroid hormone (PTH) and fibroblast growth factor 23 (FGF23). Like high blood phosphorus levels, high levels of PTH and FGF23 in the blood may also be bad for the health of your heart and blood vessels. In this study, the investigators would like to examine the effects of food additives on blood levels of phosphorus, PTH and FGF23 in individuals with normal kidney function.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, 19 - 45 years of age

Exclusion Criteria:

* abnormal urinalysis-presence of hematuria, proteinuria, or leukocyturia.
* pregnancy or breast-feeding
* Medical conditions impacting phosphate metabolism-primary hyperparathyroidism; gastrointestinal malabsorption disorders such as Crohn's Disease, ulcerative colitis, celiac disease, or liver dysfunction; hyper- or hypothyroidism; irregular menses for female subjects.
* Body Mass Index (BMI) ≥ 30 g/m2 since obesity is independently associated with impaired phosphorus metabolism.
* Medications known to affect phosphorus metabolism- current use of phosphorus supplements, high-dose or activated vitamin D compounds, regular antacid or laxative use, anticonvulsants.
* Hyper- or hypophosphatemia (≥ 4.6 mg/dl or ≤ 2.5 mg/dl respectively), hyper- or hypocalcemia (≥ 10.6 or ≤ 8.5 mg/dl respectively), or severe anemia (hemoglobin < 8 g/dl for women and < 9 g/dl for men).

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2011-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
FGF23 | 2 weeks
  Change in FGF23 levels
PTH | 2 weeks
  Change in PTH levels over 2 weeks
Serum phosphate | 2 weeks
  Change in serum phosphate over two weeks

SECONDARY OUTCOMES:
Insulin sensitivity as measured by HOMA-IR | 2 weeks
  changes in HOMA-IR over two weeks
Brachial flow mediated dilatation measured by ultrasound | 2 weeks
  change in flow mediated dilatation over two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Orlando M Gutierrez, MD, MMSc, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Gutierrez OM, Porter AK, Viggeswarapu M, Roberts JL, Beck GR Jr. Effects of phosphorus and calcium to phosphorus consumption ratio on mineral metabolism and cardiometabolic health. J Nutr Biochem. 2020 Jun;80:108374. doi: 10.1016/j.jnutbio.2020.108374. Epub 2020 Mar 19. PMID 32278118
- [Derived] Gutierrez OM, Luzuriaga-McPherson A, Lin Y, Gilbert LC, Ha SW, Beck GR Jr. Impact of Phosphorus-Based Food Additives on Bone and Mineral Metabolism. J Clin Endocrinol Metab. 2015 Nov;100(11):4264-71. doi: 10.1210/jc.2015-2279. Epub 2015 Aug 31. PMID 26323022